CLINICAL TRIAL: NCT03421197
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, 24-Week Study to Assess the Efficacy and Safety of PPC-06 (Tepilamide Fumarate) Extended Release Tablets in Subjects With Moderate-to-Severe Plaque Psoriasis (AFFIRM)
Brief Title: A Study to Assess the Efficacy and Safety of PPC-06 (Tepilamide Fumarate)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PPC-06-CD-004
Record Dates: First submitted 2018-01-23; First posted 2018-02-05 (Actual); Results first posted 2021-05-11 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — BID protein, human

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PPC-06 400 mg QD (Experimental): Tepilamide Fumarate 400 mg once per day
  Interventions: Drug: PPC-06 400 mg QD
- PPC-06 400 mg BID (Experimental): Tepilamide Fumarate 400 mg twice per day
  Interventions: Drug: PPC-06 400 mg BID
- PPC-06 600 mg BID (Experimental): Tepilamide Fumarate 600 mg twice per day
  Interventions: Drug: PPC-06 600 mg
- Placebo BID (Placebo Comparator): White placebo tablet to mimic Tepilamide Fumarate
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PPC-06 400 mg QD — Tepilamide Fumarate 400 mg tablet once per day
  Other Names: Tepilamide Fumarate 400 mg
  Arms: PPC-06 400 mg QD
Drug: PPC-06 400 mg BID — Tepilamide Fumarate tablets 400 mg twice per day
  Other Names: Tepilamide Fumarate 400 mg
  Arms: PPC-06 400 mg BID
Drug: PPC-06 600 mg — Tepilamide Fumarate tablets 600 mg twice per day
  Other Names: Tepilamide Fumarate 600 mg
  Arms: PPC-06 600 mg BID
Drug: Placebo — white tablet with no active ingredient manufactured to mimic Tepilamide Fumarate tablets
  Other Names: Placebo tablets twice per day
  Arms: Placebo BID

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter study designed to assess the safety and efficacy of PPC-06 (tepilamide fumarate) extended release in subjects with moderate-to-severe plaque psoriasis.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, placebo-controlled, multicenter study designed to assess the safety and efficacy of PPC-06 in subjects with moderate-to-severe plaque psoriasis. Study subjects will be enrolled at approximately 75 sites in the United States (US).

Approximately 400 subjects who meet the study entry criteria will be randomly assigned in a 1:1:1:1 ratio to 1 of the 4 treatment arms:

1. PPC-06 400 mg once daily (QD)
2. PPC-06 400 mg BID
3. PPC-06 600 mg BID
4. Placebo BID The maximum study duration for each subject will be approximately 29 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy males or non-pregnant females age ≥18 years at the time of screening (or who have reached the state minimum legal age of consent).
* Stable, moderate-to-severe plaque psoriasis diagnosed for at least 6 months prior to randomization (no morphology changes or significant flares of disease activity in the last 6 months in the opinion of the investigator or as reported by the subject).
* Severity of disease meeting all 3 of the following criteria prior to randomization (at the Baseline [Day 0] visit):

  1. PASI score of ≥12
  2. Total body surface area (BSA) affected by plaque psoriasis of ≥10%
  3. IGA score of >3
* Must be a candidate for phototherapy and/or systemic therapy for psoriasis.

Exclusion Criteria:

* Subjects with non-plaque psoriasis (ie, predominantly inverse, erythrodermic, predominantly guttate, or pustular psoriasis).
* Subjects with drug-induced psoriasis or subjects with drug-exacerbated psoriasis that has not resolved within 4 weeks prior to screening.
* Subjects who have received systemic non-biologic psoriasis therapy or phototherapy (including either oral and topical psoralen and ultraviolet A (PUVA) light therapy, ultraviolet B, or self-treatment with tanning beds or therapeutic sunbathing) within 4 weeks prior to the Baseline Visit.
* Subjects who had topical psoriasis treatment within the previous 2 weeks prior to the Baseline Visit.
* Subjects with history of concurrent or recent use of any biologic agent within the following washout periods prior to baseline visit:

  * Etanercept - 35 days
  * Infliximab, adalimumab - 12 weeks
  * Ustekinumab - 24 weeks
  * Any other biologic agent <5 half-lives prior to the Baseline Visit
* Subjects with history of use of any investigational drug within 28 days prior to randomization, or 5 pharmacokinetic/ pharmacodynamic half-lives (whichever is longer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Sidgiddi, MD, Study Director — Dr. Reddy's Laboratories, Inc
Locations (74):
- United States (74):
  - Site 144, Glendale, Arizona
  - Site 167, Phoenix, Arizona
  - Site 158, Phoenix, Arizona
  - Site 170, Tempe, Arizona
  - Site 157, Bryant, Arkansas
  - Site 125, Rogers, Arkansas
  - Site 133, Fountain Valley, California
  - Site 107, Fremont, California
  - Site 121, Fresno, California
  - Site 153, Fullerton, California
  - Site 176, Los Angeles, California
  - Site 178, Los Angeles, California
  - Site 182, Los Angeles, California
  - Site 156, Murrieta, California
  - Site 141, San Diego, California
  - Site 155, Santa Rosa, California
  - Site 137, Clearwater, Florida
  - Site 130, Coral Gables, Florida
  - Site 143, Hialeah, Florida
  - Site 145, Hialeah, Florida
  - Site 181, Hialeah, Florida
  - Site 149, Miami, Florida
  - Site 105, Miami, Florida
  - Site 174, Miami, Florida
  - Site 164, Miami, Florida
  - Site 123, Miami, Florida
  - Site 112, Miramar, Florida
  - Site 172, New Port Richey, Florida
  - Site 152, Orange Park, Florida
  - Site 154, Pembroke Pines, Florida
  - Site 110, Sweetwater, Florida
  - Site 150, Tampa, Florida
  - Site 113, Tampa, Florida
  - Site 132, Marietta, Georgia
  - Site 124, Savannah, Georgia
  - Site 122, Nampa, Idaho
  - Site 179, Wheaton, Illinois
  - Site 115, Indianapolis, Indiana
  - Site 171, New Albany, Indiana
  - Site 139, Overland Park, Kansas
  - Site 165, Louisville, Kentucky
  - Site 131, Louisville, Kentucky
  - Site 142, Louisville, Kentucky
  - Site 119, Baton Rouge, Louisiana
  - Site 126, New Orleans, Louisiana
  - Site 128, Clinton Township, Michigan
  - Site 129, Fridley, Minnesota
  - Site 111, Kansas City, Missouri
  - Site 109, Omaha, Nebraska
  - Site 127, Las Vegas, Nevada
  - Site 180-, Las Vegas, Nevada
  - Site 103, New York, New York
  - Site 177, New York, New York
  - Site 104, New York, New York
  - Site 161, Rochester, New York
  - Site 146, Stony Brook, New York
  - Site 108, High Point, North Carolina
  - Site 116, Wilmington, North Carolina
  - Site 118, Beachwood, Ohio
  - Site 169, Cincinnati, Ohio
  - Site 114, Johnston, Rhode Island
  - Site 134, Mt. Pleasant, South Carolina
  - Site 100, Rapid City, South Dakota
  - Site 148, Austin, Texas
  - Site 160, Bellaire, Texas
  - Site 162, Houston, Texas
  - Site 102, Houston, Texas
  - Site 106, San Antonio, Texas
  - Site 101, San Antonio, Texas
  - Site 159, Sugar Land, Texas
  - Site 136, Orem, Utah
  - Site 166, Norfolk, Virginia
  - Site 135, Burien, Washington
  - Site 147, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PPC-06 400 mg QD | PPC-06 400 mg BID | PPC-06 600 mg BID | Placebo BID
Started | 105 | 107 | 107 | 107
Completed | 67 | 68 | 56 | 62
Not Completed | 38 | 39 | 51 | 45

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PPC-06 400 mg QD | PPC-06 400 mg BID | PPC-06 600 mg BID | Placebo BID | Total
Number analyzed (Participants) | 105 | 107 | 107 | 107 | 426
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (13.18) | 51.0 (12.29) | 50.2 (13.74) | 49.3 (12.59) | 49.6 (12.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 43 | 43 | 43 | 169
  Male | 65 | 64 | 64 | 64 | 257
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 0 | 1 | 4
  Asian | 1 | 3 | 2 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 6 | 4 | 11 | 5 | 26
  White | 97 | 96 | 92 | 97 | 382
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 2 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 105 | 107 | 107 | 107 | 426
Psoriasis Area and Severity Index (PASI) [Mean (Standard Deviation); unit: units on a scale] — The PASI is a measure of the average redness, thickness, and scaliness of the lesions (each graded on a 0-4 scale) and is weighted by the area of involvement. The three signs are assessed on 4 body regions - Head, Trunk, Upper Limbs and Lower Limbs. Scores for each sign are assigned on all body regions and calculated per a validated formula. The minimum possible score is 0, while maximum score on this scale is 72. A higher PASI at baseline indicates greater disease severity.
  units on a scale | 18.41 (6.377) | 18.56 (8.004) | 18.00 (6.680) | 17.26 (6.169) | 18.05 (6.842)

OUTCOME MEASURES:

1. Primary Outcome: Achieving Psoriasis Area and Severity Index (PASI) - 75 at the End of Week 24
Description: The percentage of subjects who achieve a reduction of 75% or greater from Baseline in the Psoriasis Area and Severity Index (PASI-75) The PASI is a measure of the average redness, thickness, and scaliness of the lesions (each graded on a 0-4 scale) and is weighted by the area of involvement. The minimum possible score on this scale is '0', while the maximum score on this scale is 72. A lower score on this scale at the end of the study indicates an improvement in the condition of subject.
Time Frame: End of Week 24
Population: Full Analysis Set (FAS) Population which included all randomized subjects who received at least one dose of IP and had at least one post-dose efficacy assessment.
Measure: Number; unit: percentage of total participants
Arm/Group | PPC-06 400 mg QD | PPC-06 400 mg BID | PPC-06 600 mg BID | Placebo BID
Number analyzed (Participants) | 101 | 102 | 101 | 102
percentage of total participants | 39.7 | 47.2 | 44.3 | 20.0

2. Primary Outcome: Achieving the Investigator's Global Assessment (IGA) Score of 0 or 1
Description: The Percentage of subjects who achieve the Investigator's Global Assessment (IGA) score of clear or almost clear (IGA score 0 or 1)
  Score Grade Definition 0 Clear: No signs of psoriasis
  1. Almost clear: No thickening to minimal plaque elevation; Normal to slight pink coloration/faint erythema; Focal to minimal scaling
  2. Mild: Slight elevation/thickening; Pink to light red coloration; Predominantly fine scaling partially or mostly covering lesions
  3. Moderate: Clearly distinguishable/distinct thickening; Definite red coloration; Coarse scaling covering most plaques
  4. Severe: Marked thickening with hard/sharp edges; Bright to deep dark red coloration; Thick/coarse scaling covering almost all or all lesions
  A lower score on this scale at the end of the study indicates an improvement in the disease condition.
Time Frame: End of Week 24
Population: Full Analysis Set (FAS) Population included all randomized subjects who received at least one dose of IP and had at least one post-dose efficacy assessment.
Measure: Number; unit: percentage of total participants
Arm/Group | PPC-06 400 mg QD | PPC-06 400 mg BID | PPC-06 600 mg BID | Placebo BID
Number analyzed (Participants) | 101 | 102 | 101 | 102
percentage of total participants | 35.7 | 41.4 | 44.4 | 22.0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of signing the informed consent, up to 30 days after the last dose.
Description: Adverse events were assessed at all study visits. Adverse events were monitored by the investigator from the time of signing informed consent, up to 30 days after the subject has stopped study treatment or until the AE had resolved or stabilized.
  Adverse events were evaluated in the Safety Population.
Arm/Group | PPC-06 400 mg QD | PPC-06 400 mg BID | PPC-06 600 mg BID | Placebo BID
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/107 | 0/106 | 0/107
Serious Adverse Events (participants affected / at risk) | 3/105 | 3/107 | 0/106 | 2/107
Other Adverse Events (participants affected / at risk) | 30/105 | 42/107 | 68/106 | 9/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PPC-06 400 mg QD (N=105) | PPC-06 400 mg BID (N=107) | PPC-06 600 mg BID (N=106) | Placebo BID (N=107)
Dyspnoea/Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Allergic Reaction
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Right femur
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — C-Spine Compression
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Staphylococcal skin infection in right lower leg
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PPC-06 400 mg QD (N=105) | PPC-06 400 mg BID (N=107) | PPC-06 600 mg BID (N=106) | Placebo BID (N=107)
Lymphopenia (Blood and lymphatic system disorders) | 4 (4) | 4 (5) | 10 (10) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 5 (5) | 6 (7) | 5 (5) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 7 (12) | 19 (20) | 24 (32) | 5 (5)
Nausea (Gastrointestinal disorders) | 7 (8) | 7 (7) | 11 (11) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 4 (4) | 5 (6) | 12 (13) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 1 (1) | 6 (7) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-26): https://cdn.clinicaltrials.gov/large-docs/97/NCT03421197/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/97/NCT03421197/SAP_001.pdf